CLINICAL TRIAL: NCT04015284
Title: Intraoperative Pain and Quality of the Surgical Nerve Block During Arthroscopic Shoulder Surgery Assessed by the NOL Index When Comparing the Combined Suprascapular and Posterior Cord Nerve Blocks to the Interscalene Brachial Plexus Block
Brief Title: Intraoperative Pain and Quality of Surgical Block During Shoulder Surgery Assessed by NOL Index
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This type of surgery is no longer done at HMR, relocated to other centers
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, MD, PhD, Professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-1743
Record Dates: First submitted 2019-04-08; First posted 2019-07-10 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Shoulder Surgery; Regional Anesthesia Morbidity
Keywords: NOL monitoring; regional anesthesia; interscalene brachial plexus block; shoulder arthroscopy

STUDY DESIGN:
Intervention Model Description: 2 groups of patients. Randomization into groups SSNP + PCB or ISBPB as per randomization list, for a total of 100 patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSNB + PCB (Experimental): Single shot US-guided suprascapular nerve block (SSNB) with 5 mL ropivacaine 0.5%, then single shot US-guided posterior cord block (PCB) with 10 ml ropivacaine 0.5%.
  Interventions: Procedure: Suprascapular Nerve Block + Posterior Cord Block
- ISBPB (Active Comparator): Single shot US-guided interscalene brachial plexus block (ISBPB) with 15 mL ropivacaine 0.5%.
  Interventions: Procedure: Interscalene Brachial Plexus Block

INTERVENTIONS:
Procedure: Suprascapular Nerve Block + Posterior Cord Block — The patient lies supine with the head turned to the contralateral side to the block. Using a linear high-frequency ultrasound probe, the proximal suprascapular nerve is visualized before it turns toward the suprascapular notch. It is blocked using 5mL of ropivicaine 0.5%. The posterior cord is readily visualized when performing an infraclavicular brachial plexus block. It is blocked using 10mL of ropivicaine 0.5%.
  Other Names: SSNB+PCB
  Arms: SSNB + PCB
Procedure: Interscalene Brachial Plexus Block — The patient lies supine with the head turned to the contralateral side to the block. Using a linear high-frequency ultrasound probe, the interscalene groove is visualized along with the roots of the brachial plexus. The block is performed with 15mL of ropivacaine 0.5%.
  Other Names: ISPB
  Arms: ISBPB

SUMMARY:
Postoperative analgesia for shoulder surgery is typically achieved by providing an interscalene brachial plexus block. However, a very common side effect of this block is hemi-diaphragmatic paralysis, a state which may not be tolerated in patients with pulmonary conditions such as COPD. Recently, clinicians have explored new ways to provide satisfactory analgesia while minimizing the pulmonary side effects of the interscalene nerve block. One of these solutions might be to offer the patient a suprascapular nerve block combined to a posterior cord block. Since these blocks are performed lower in the neck or under the clavicle, the phrenic nerve is less likely to be blocked. Thus, fewer respiratory side effects have been reported when using such blocks. This prospective observational study will evaluate the NOL response to surgical stimuli and the opioid requirements intraoperatively in patients undergoing shoulder arthroscopies with either a supraclavicular and posterior cord blocks or an interscalene block.

Study Design: Prospective, randomized open label non-inferiority trial. Subject Population: Adults scheduled to undergo elective shoulder arthroscopy Sample Size: 100 patients Study Duration: Starts February 2019 - Ends February 2021 - Interim analysis at 50 patients Study Center: Maisonneuve-Rosemont Hospital, CEMTL, Montreal, Quebec, Canada

DETAILED DESCRIPTION:
The main hypothesis of this study is that the suprascapular block combined with a posterior cord block is not inferior to the interscalene brachial plexus block in terms of intraoperative analgesia. We postulate that intraoperative opioid requirements will not differ significantly in patients who receive either block.

Our secondary objectives will consist in looking at the differences in intraoperative anesthetic consumption, NOL index alterations, postoperative opioid consumption, pain scores, arm motor block, diaphragmatic paresis, patient satisfaction and time for readiness to discharge from PACU. We hypothesize that these outcomes will be similar in both groups, with the exception of a potential reduction in arm motor block and diaphragmatic paresis in the combined suprascapular and posterior cord block group.

After having obtained institutional ethics board approval of the study, patients older than 18 years old, scheduled for a first elective shoulder arthroscopy under general anesthesia will be screened in the pre-anesthesia clinic. They will be approached and the whole study procedures will be explained extensively. Interested patients will be invited to sign the consent form (see appendix). Patients will have the right to opt out at any time. The investigators will meet the patients again on the morning of the surgery to address any concerns. After consent, a study number will be allocated to the patient in ascending order.

Two groups will be evaluated:

* Group A: single shot US-guided suprascapular nerve block with 5 mL ropivacaine 0.5%, then single shot US-guided posterior cord block with 10 ml ropivacaine 0.5%.
* Group B: single shot US-guided interscalene brachial plexus block with 15 mL ropivacaine 0.5%.

Tests will be done to evaluate the nerve block-induced loss of sensation to ice prior to entering the operating room (OR). Diaphragmatic excursion will be evaluated using an abdominal curvilinear ultrasound probe, and will be classified as being normal, paradoxical or immobile. Normal motion is caudad movement during inspiration. Paradoxical motion is cephalad movement during inspiration.

Once in the operating room, all routine monitors are connected. Moreover, the PMD TM monitor as well as the BIS® monitor are connected to the anesthesia machine and to the patient. Both study monitors are switched on and will record their respective indices continuously for the duration of the anesthesia. General anesthesia will be induced with propofol (1-2 mg/kg IV; Pharmascience Inc, Canada), remifentanil (1 µg/kg IV bolus; Teva, Canada) and rocuronium (0.6-1 mg/kg IV; Sandoz Canada Inc). A bolus of dexamethasone 4mg IV will be administered after induction of general anesthesia.

Patients will also have received oral acetaminophen 1g and celecoxib 400 mg preoperatively. Intubation with an endotracheal tube is performed once the patient is adequately paralyzed (no responses to the TOF stimulation). All drugs are given according to the adjusted body weight of the patient. This is calculated with Robinson's formula: where TBW is total body weight and IBW is ideal body weight (21-22). Immediately after intubation, anesthesia is maintained with desflurane while targeting a BIS value between 45 and 55, and a remifentanil infusion and boluses are used for a NOL below 25. At the end of anesthesia, when the surgeon starts closing the wounds, an IV bolus of hydromorphone 7 mcg/kg of adjusted body weight is administered. The remifentanil infusion and desflurane are discontinued when dressing starts. Emergence and extubation are done in the OR. All times (start skin closure, start dressing, stop desflurane and remifentanil) will be precisely reported in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1,2,3.
* Age 18 years or older
* Elective shoulder arthroscopic surgery under general anesthesia and nerve block performed preoperatively

Exclusion Criteria:

* Serious cardiac arrhythmias (including atrial fibrillation) or unstable coronary artery disease.
* Coagulation disorders.
* Patient refusal.
* Anatomical disorders and/or neuropathic disease.
* BMI above 40.
* History of substance abuse.
* Chronic use of psychotropic and/or opioid.
* History of psychiatric diseases needing treatment.
* Contraindications to nerve block for shoulder surgery.
* Allergy to remifentanil or any drug in the study protocol.
* Failure of nerve block performed in the preoperative block room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Dose of remifentanil in mcg/kg/h during the surgery period | Intraoperative from incision until wound dressing
  The main criterion will be evaluating the dose of remifentanil per kg per hour of surgery needed intraoperatively to keep a NOL index below the threshold of 25.

SECONDARY OUTCOMES:
NOL response after surgical incisions (area under curve) | Intraoperative
  NOL response after surgical incisions 1 (located 2 cm inferior and 1 cm medial to posterolateral corner of acromion) of the shoulder (by calculating the area under the curve of NOL for the 5 minutes following incision 1).
NOL response after surgical incisions (area under curve) | Intraoperative
  NOL response after surgical incisions 2 (located slightly inferior to coracoid) of the shoulder (by calculating the area under the curve of NOL for the 5 minutes following incision 1).
Total dose remifentanil in mcg | Intraoperative
  Total dose of remifentanil in mcg from incision until wound dressing
Number of remifentanil boluses (n) | Intraoperative
  Number of remifentanil boluses administered to the patient from incision until wound dressing
Desflurance consumption in ml | Intraoperative from incision until wound dressing
  Intraoperative consumption of desflurane in mL
Time to awakening in minutes | Intraoperative
  Time to awakening in minutes.
Time to extubation in minutes | Intraoperative
  Time to extubation in minutes.
PACU pain scores on a scale from 0 to 10 | From entrance in PACU until PACU discharge e.g. up to 3 hours after surgery maximum
  PACU pain scores
Grip strength in mmHg | in PACU e.g. up to 3 hours after surgery maximum
  Grip strength before nerve blockade and prior to PACU discharge, as measured in mmHg by a pressure transducer connected to a 1000mL saline bag.
Diaphragmatic paresis induced by the nerve block by ultrasound | 30 minutes after nerve block and before general anesthesia and surgery, in awake patient
  Ipsilateral diaphragmatic excursion 30 minutes after block completion (normal, paradoxical or no movement).
Patient dyspnea on a scale from 0 to 10 | PACU e.g. up to 3 hours after surgery maximum
  Patient dyspnea prior to PACU discharge on a scale from 0 to 10.
Time to readiness for discharge from PACU in minutes | PACU e.g. up to 3 hours after surgery maximum
  Time to readiness for discharge from PACU = time in minutes to reach an Aldrete score at 9 for discharge
24h pain scores on a scale from 0 to 10 at rest | Postoperative at H24, 24 hours after surgery
  24h pain scores, H24
48h pain scores on a scale from 0 to 10 at rest | Postoperative at H48, 48 hours after surgery
  48h pain scores
24h pain scores on a scale from 0 to 10 during mobilization | Postoperative at H24, 24 hours after surgery
  24h pain scores during mobilization
Per os postoperative (after PACU discharge) morphine equivalent consumption in mg at 8, 16, 24, 32, 40, 48 hs postoperatively | Postoperative for 2 days 48 hours after surgery
  Per os opioid consumption in mg of equivalent morphine (every 8 hours by nurses or with a diary in patients with same day surgery).
Duration of motor block in minutes strength | Postoperative for day 1 H24 24hours after surgery
  Duration of motor block in minutes, as measured by time to return of normal grip strength.
Patient satisfaction on a scale from 0 to 100 | Postoperative at 24h, 24 hours after surgery
  Patient satisfaction at 24 hours on a scale from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebe, MD, PhD, Principal Investigator — CIUSSS de l'Est de Montreal
Locations (1):
- Hôpital Maisonneuve-Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal, Quebec, Canada